CLINICAL TRIAL: NCT05506735
Title: The Role of the Seven Sweeps in the Prevention of the Prostate Cancer Among Those With a Positive Family History: A Retrospective Cohort Study
Brief Title: The Role of the Seven Sweeps in the Prevention of the Prostate Cancer Among Those With a Positive Family History
Acronym: PSA
Status: Completed | Type: Observational
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hashim Talib Hashim, Doctor (MBChB), University of Baghdad
Other Study IDs: 003
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer; Prostatic Neoplasms; Prostatic Hyperplasia
Keywords: Prostate cancer; Prostate hyperplasia; The seven sweeps
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The seven sweeps is a recommended act performed by men after urinating in order to be confident that no urine is left in the urethra, and its not compulsory to perform. It is performed by the following way: after urinating, the anus is first purified if it has become impure; then, the middle finger of the left hand is slid three times from the anus up to the scrotum; then, the thumb is placed on the penis and the forefinger is placed under the penis, and the thumb and forefinger are pulled three times along the penis up to the point of circumcision; finally, the end of the penis is pressed three times.

DETAILED DESCRIPTION:
The investigators have investigated 350 people who have been doing this habit for at least 20 years of their life and they have a family history of prostatic cancer to check the effect of this procedure on the prevention of the cancer. The investigators have excluded 135 participants of them because they have not full-filled the criteria of inclusion. So 215 of them have been included and investigated using PSA and prostate ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Family history of prostate cancer, more than 40 years of age, is doing the seven sweeps habit for at least 20 years, has not any urinary problems or chronic diseases.

Exclusion Criteria:

* No family history of prostate cancer, less than 40 years of age of more than 70 years old, has a urinary problem or chronic diseases.

Ages: 40 Years to 70 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Any human with prostate organ who identified himself as a man and he has a male genital organs of penis and testes.
Study Population: We included 350 participants and 135 if them were excluded. Only 215 who full-filled the criteria were included.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Prostate specific antigen | 30 minutes
  PSA is a protein made by the prostate gland. The amount of PSA may be higher in men who have prostate cancer, benign prostatic hyperplasia (BPH), or infection or inflammation of the prostate. Also called prostate-specific antigen test.

SECONDARY OUTCOMES:
Prostate ultrasound | 30 minutes
  Using the sonography to locate and measure the thickness and the tissue of the prostate.

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Talib T Hashim, MBChB, Principal Investigator — University of Baghdad, College of Medicine
Locations (1):
- Al-Dar medical Center, Nasiriyah, Thi Qar, Iraq